CLINICAL TRIAL: NCT03268980
Title: Study of Smoking Prevalence at the "Hospices Civils de Lyon"
Brief Title: Smoking Prevalence at a University Hospital
Acronym: TABAC-HCL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0481
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2017-08

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients group: All patients (over 18y) admitted to the Hospices Civils de Lyon the day of the study, whatever the reason, able to fullfill the questionnaire by themselves.
  Interventions: Other: Questionnaire students and patients group
- Hospital staff group: Anyone, whatever age and trade, paid directly by the Hospices Civils de Lyon on the day of the survey, regardless of the duration of the employment contract, and present on one of the sites of the Hospices Civils de Lyon the day of the investigation.
  Interventions: Other: Questionnaire Hospital Staff group
- Students group: Everyone who is regularly enrolled in one of the schools or institutes of the Hospices Civils de Lyon or in one of the two faculties of medicine of the Université Lyon I, in any initial training and present on one of the sites of the faculties the day of the investigation
  Interventions: Other: Questionnaire students and patients group

INTERVENTIONS:
Other: Questionnaire Hospital Staff group — One-page questionnaire with 15 questions about tobacco habits
  Groups: Hospital staff group
Other: Questionnaire students and patients group — One-page questionnaire with 17 questions about tobacco habits
  Groups: Patients group; Students group

SUMMARY:
* Tobacco is the leading risk factor for avoidable mortality in France and around the world. It is also the second cause of life with disability in the world and the leading preventable risk factor for cancer in France and worldwide.
* The "Health Barometer" studies carried out for 25 years in France by Santé-Publique France assessed prevalence of smoking in the lay population. These studies showed that smoking prevalence has stabilized among 15-75 year olds (34.1% of current smokers) with a slight decrease in regular smoking (from 29.1% in 2010 to 28.2% in 2014).
* Data on the prevalence of smoking among hospital staff are contradictory. Some studies find a higher prevalence of active smoking than the general population; others have a lower prevalence. However, it appears that an active prevention policy with hospital staff can significantly and rapidly reduce the prevalence of active smoking.
* The prevalence of active smoking in patients is logically higher than in the general population (at comparable age).
* The data on the prevalence of smoking among medical students are also contradictory. Yet, this population is a special interest group given their future investment in patient care.
* Cannabis use also appears to be an independent risk factor for respiratory diseases and broncho-pulmonary cancers. Cannabis use among health students is not uncommon (11.5% of students). To our knowledge, the measurement of the prevalence of Cannabis use in an all-patient population of a hospital-university facility has never been achieved.
* According to the health barometer 2014, about a quarter of 15-75 year olds have already tried electronic cigarettes and 6% are regular current users. Although the toxicity of the electronic cigarette and its interest in weaning remain controversial, its use to patients, staff or patients has been reported very little.

The aim of this study is to assess the impact of collective and individual tobacco control measures by measuring the prevalence of smoking on a given day at the "Hospices Civils de Lyon", among patients, staff and students present on a given day.

ELIGIBILITY:
Inclusion Criteria:

- Patients group: Any person, over 18 years of age, hospitalized in one of the establishments of the Hospices Civils de Lyon, whatever the reason and the duration.

- Hospital staff group: Anyone, whatever age and trade, paid directly by the Hospices Civils de Lyon on the day of the survey, regardless of the duration of the employment contract, and present on one of the sites of the Hospices Civils de Lyon the day of the investigation.

- Students group: Everyone who is regularly enrolled in one of the schools or institutes of the Hospices Civils de Lyon or in one of the two faculties of medicine of the Université Lyon I, in any initial training and present on one of the sites of the faculties the day of the investigation

Exclusion Criteria:

* Patients group:

  * Refusal to participate
  * Refusal of parents or legal representative for minors or adults of full age.
  * Child under the age of 18 at the time of the survey.
  * Individual who do not speak, understand or read the French language.
  * Non-hospitalized individuals (including external consultants).
  * Patient whose clinical status is not compatible with the administration of the questionnaire (eg, disorders of consciousness, severe cognitive impairment, severe speech disturbances, extreme asthenia) as judged by the service health framework and / or the medical team of the service.
  * Individual currently incarcerated.
* Hospital staff group:

  * Refusal to participate.
  * Temporary staff (not paid directly by the Hospices Civils de Lyon on the day of the survey).
  * Students present on the day of the survey, and in particular: hospital students, nursing students and nursing assistants.
* Students group:

  * Refusal to participate
  * Professional present in the school / institute / faculty as part of continuing education.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three populations are identified:
  * Patients group: All persons admitted to the Hospices Cvils de Lyon on the day of the investigation, whatever the reason.
  * Hospital staff group: All members of the staff of the Hospices Civils de Lyon, present at their place of work on the day of the inquiry, whatever their status.
  * Students group: All students of the faculties of medicine of Université Lyon I and of the Hospices Civils de Lyon training institutes present in the university or training institute on the day of the survey, whatever their status.
Sampling Method: Non-Probability Sample
Enrollment: 11276 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Measure the prevalence of smoking one day given to the Hospices Civils de Lyon, in patients, the members of the staff and students present one day | One day
  The aim of this study is to determine the proportion of active smoker / smoker weaned / non-smoker in each group (patients / hospital staff / students).
  Data are collected by a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie Aigue Spécialisée et Cancérologie Thoracique - Hôpital Lyon-Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No